CLINICAL TRIAL: NCT01264120
Title: The Impact of a Bariatric Rehabilitation Service on Weight Loss and Psychological Adjustment.
Brief Title: The Impact of a Bariatric Rehabilitation Service on Patient Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Surrey (Other)
Collaborators: Western Sussex Hospitals NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PB-PG-0909-20178 NIHR
Record Dates: First submitted 2010-12-16; First posted 2010-12-21 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: Obesity; Bariatric surgery; Health Psychology
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Psychology Intervention (Experimental): A 50 minute health psychology behavioural intervention with sessions pre-surgery, post-surgery and at 3 month follow up.
  Interventions: Behavioral: Health Psychology Intervention
- Control Group (No Intervention): The control group receive usual care through the bariatric surgery process.

INTERVENTIONS:
Behavioral: Health Psychology Intervention — The health psychology intervention will involve a bariatric rehabilitation service (BRS) which will involve those allocated to the intervention receiving usual care plus three 50 minute sessions with a health psychologist pre-operatively (1 week before surgery), perioperatively (before they are discharged from hospital) and at 3 month follow up.
  Other Names: Bariatric rehabilitation
  Arms: Health Psychology Intervention

SUMMARY:
Obesity is a major health problem that is affecting more and more people's lives. One of the most successful treatments for obesity is weight loss surgery. Not all patients, however, lose the desired amount of weight, some regain weight and some have the surgery reversed. Interviews with patients and discussions with patient support groups indicate that many of the 'unsuccessful' patients feel unprepared for the operation and describe how although the surgery fixes their body it neglects their mind. They would therefore like to have more psychological support.

The present study aims to set up and evaluate a health psychology led bariatric rehabilitation service (BRS) and determine the impact of such a service on patient outcomes following surgery. The BRS would offer information, support and mentoring pre and post surgery and address psychological issues such as dietary control, self esteem, coping and emotional eating. It is predicted that a bariatric rehabilitation service would primarily improve weight loss following surgery but would also aid changes in other aspects of the patient's well being.

Obesity is a risk factor for a multitude of illnesses such as heart disease, diabetes and cancer. If effective, obesity surgery improves a patient's health and reduces their need for NHS care. If unsuccessful then the costs include not only subsequent NHS costs due to these other illnesses but also the costs of the unsuccessful operation and the emotional cost to the patient. The bariatric rehabilitation service should help to improve the effectiveness of surgery which in the longer term is likely to be cost effective.

This research is a direct response to the needs identified by patients and by offering a more comprehensive bariatric service the success and subsequent health and well being of obese patients should be improved.

DETAILED DESCRIPTION:
Design: The study will involve a trial (open randomised parallel group control trial) with patients allocated to receive either usual care or the bariatric rehabilitation service (BRS) pre and post bariatric (obesity) surgery. Follow up measures will be recorded at 3, 6 and 12 months post-surgery at routine follow-up clinics. In addition, qualitative interviews will be carried out with 20 participants from both arms of the trial (BRS n=10; usual care n=10).

Piloting: The contents of the bariatric service and the follow up measures are based on pilot work. This pilot work has already been completed exploring what bariatric patients want and why bariatric surgery either fails or succeeds from the patients' perspective. Furthermore, pilot research has explored the impact of bariatric surgery on changes in mood, cognitions and eating behaviours. The quantitative measures and qualitative responses derived from these studies will form the basis of the intervention and the measures for the present study.

Sample: St Richard's Hospital in Chichester, West Sussex offers a NHS based bariatric service for obese patients with a BMI over 40 (or 35 with serious co morbidities). This is the largest centre in the UK, with 600 patients per year receiving a bariatric operation at this clinic (70% being a primary bypass and 20% bands (the remaining 10% are revisions)). Patients will be recruited if they have been approved for surgery and had their date set for their operation. The consultant surgeon, Mr Chris Pring is a collaborator on this proposal.

Procedure: Ethical approval will be in place before the start of the project. In the week before their operation patients attend the bariatric clinic for routine tests. When patients are sent their appointment letters they will be sent the information sheet along with it to give them approximately 2 weeks to think about whether they would like to take part. At the appointment patients will see the researcher who will explain the trial, obtain consent and randomly allocate the patient to either the usual care condition or the bariatric rehabilitation service (BRS) condition.

Randomisation: All patients who fulfil the inclusion criteria will be approached by the researcher, asked to read an information sheet and if interested offered a written consent form. Once a patient is consented the researcher will contact the clinical trial unit at Surrey University who will provide third party blinded randomization to either the BRS or usual care.

Timeline: The study will take 34 months. New patients will be recruited over a 12 month period and followed up for 12 months postoperatively. The first 6 months will involve preparation, setting up procedures for data collection and training the health psychologist. The next 25 months will involve rolling out the intervention, recruitment, randomly allocating patients to the 2 conditions, providing the BRS and collecting data on the evaluation of service. At 18 months the 20 interviews will take place and be transcribed. The final 3 months will be spent analyzing the data, assessing cost-effectiveness, disseminating the results to patients and health professionals and writing up findings for publication.

ELIGIBILITY:
Inclusion Criteria:

* if they consent
* aged 18 or over
* have attended the bariatric clinic at Chichester
* been accepted for surgery
* have funding in place for surgery (i.e. their primary care trust has agreed to pay for their surgery).

Exclusion Criteria:

* those who do not wish to take part in the randomisation
* those who do not wish to take part in the intervention
* those who will not be having bariatric surgery because they are not a suitable patient
* those who will not be having bariatric surgery because they can not secure funding from their primary care trust for the surgery
* those who cannot effectively read or speak English, as this would pose a difficulty in implementing the intervention and for data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in weight and BMI | Baseline, 3, 6 and 12 months
  The weight and height of patients will be obtained to determine BMI change over the duration of the intervention.

SECONDARY OUTCOMES:
Change in psychological measures | Baseline, 3,6 and 12 months.
  The secondary outcome measure is the impact of the BRS on patients' quality of life, dietary control, coping strategies and emotional eating.
Cost-effectiveness | At the end of the intervention
  The cost-effectiveness of the intervention will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ogden, PhD, Principal Investigator — University of Surrey
Locations (1):
- St Richards Hospital, Chichester, West Sussex, United Kingdom

REFERENCES:
- [Background] Hollywood A, Ogden J, Pring C. The impact of a bariatric rehabilitation service on weight loss and psychological adjustment--study protocol. BMC Public Health. 2012 Apr 5;12:275. doi: 10.1186/1471-2458-12-275. PMID 22480247
- [Derived] Ogden J, Hollywood A, Pring C. The impact of psychological support on weight loss post weight loss surgery: a randomised control trial. Obes Surg. 2015 Mar;25(3):500-5. doi: 10.1007/s11695-014-1428-2. PMID 25200170